CLINICAL TRIAL: NCT05187845
Title: Geriatrisch-Onkologische Studie Zur Lebensqualität Und Selbstständigkeit Nach Radiotherapie Geriatric-oncological Study on Quality of Life and Independence After Radiotherapy
Brief Title: Geriatric-oncological Study on Quality of Life and Independence After Radiotherapy
Acronym: GOLD-I
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department Director, University Hospital Heidelberg
Other Study IDs: RadOnk_2021_GOLD-I
Record Dates: First submitted 2021-12-21; First posted 2022-01-12 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Age <70
Keywords: quality of life after radiotherapy; independence after radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elderly patients * with multiple comorbidities are underrepresented in most radio-oncology studies. In times of individualized therapy and when weighing up oncological over- or under-therapy, this observational study is a step towards the implementation of established geriatric instruments and concepts in radiation oncology. As part of the initial outpatient consultation on radiotherapy, the quality of life of patients older than 70 years before the start of therapy is assessed using the EORTC QLQ-C30 and ELD14 questionnaires. Furthermore, a geriatric screening is carried out using the G8 questionnaire. The geriatric screening carried out in routine clinical practice with little effort is used to filter out patients with no risk of increased vulnerability - these participants do not require any further examinations.

DETAILED DESCRIPTION:
Vulnerable patients with deficits (G8 score <15 pts) receive a geriatric assessment (Comprehensive geriatric assessment (CGA)) consisting of abbreviated comprehensive geriatric assessment (aCGA), appetite (Mini Nutritional Assessment (short form = MNA-SF)) at the beginning and end of radiotherapy ), physical functionality (Short physical performance battery) and measurement of hand strength. In addition, these patients receive an individualized inpatient geriatric-oncological complex treatment, which is already implemented analogous to the palliative complex treatment. The patients receive targeted support from trained nursing staff, social services, physiotherapy, nutritional advice, hospital pharmacies and psycho-oncology. At the end of the oncological therapy and for the first aftercare after the end of therapy, the questionnaires on quality of life are filled out again in order to analyze changes. Initially, 20 patients are to be treated in a first phase (feasibility) in this concept of geriatric-oncological complex treatment in order to build up and expand the necessary structures for an interdisciplinary complex treatment and to set parameters for adherence to the therapy concept and maintaining quality of life and independence in the activities of the daily life for this collective of patients. As part of a follow-up study, vulnerable patients are then to be stratified and randomized using these parameters so that a more detailed analysis is possible.

ELIGIBILITY:
Inclusion Criteria:

* Age from 75 years
* G8-Screening <15Pkt
* Potentially curative radiotherapy

Exclusion Criteria:

* no written informed consent
* life expectancy< 6 month

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 20 patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Radiation associated changes in the independence in the activities of daily living | upt to 6 month after radiotherapy
  Changes in the Barthel Index
Compliance to radiotherapy treatment | through treatment time of radiotherapy, an average of 6 weeks
  number of Events of premature termination of planned radiotherapy treatment

SECONDARY OUTCOMES:
Therapy associated toxicity | up to 6 month after radiotherapy
  Changes in toxicity assesment according to CTC
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  Sex
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  age
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  Barthel Index
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  Tumor entitiy
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  type of Radiation treatment
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  time of radiation treatment
Analysis of prognostic factors for radiotherapy Treatment success | during radiotherapy
  rate of hospitalization Events
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  rate of hospitalization events
Analysis of prognostic factors for radiotherapy Treatment success | up to 6 month after radiotherapy
  required medications

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, Prof, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany